CLINICAL TRIAL: NCT03241459
Title: Randomized & Controlled Noninferiority Trial to Evaluate Safety & Clinical Efficacy of SurVeil™ Drug-Coated Balloon (DCB) iN Treatment of Subjects With Stenotic Lesions of Femoropopliteal Artery Compared to Medtronic IN.PACT® Admiral® DCB
Brief Title: Safety and Efficacy of the SurVeil™ Drug-Coated Balloon
Acronym: TRANSCEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SurModics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUR17-001
Record Dates: First submitted 2017-08-01; First posted 2017-08-07 (Actual); Results first posted 2024-04-09 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease; Artery Disease, Peripheral; Femoropopliteal Artery Occlusion
Keywords: Percutaneous Transluminal Angioplasty; PTA; Peripheral Artery Disease; PAD; Paclitaxel
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Surmodics SurVeil DCB (Experimental): Surmodics SurVeil Drug-Coated Balloon is an investigational device coated with paclitaxel.
  Interventions: Device: Surmodics SurVeil DCB
- Medtronic IN.PACT Admiral DCB (Active Comparator): Angioplasty procedure with a paclitaxel-coated, percutaneous transluminal angioplasty (PTA) balloon catheter.
  Interventions: Device: Medtronic IN.PACT Admiral DCB

INTERVENTIONS:
Device: Surmodics SurVeil DCB — Angioplasty procedure with a paclitaxel-coated, percutaneous transluminal angioplasty (PTA) balloon catheter.
  Arms: Surmodics SurVeil DCB
Device: Medtronic IN.PACT Admiral DCB — Angioplasty procedure with a paclitaxel-coated, percutaneous transluminal angioplasty (PTA) balloon catheter.
  Arms: Medtronic IN.PACT Admiral DCB

SUMMARY:
To demonstrate the safety and efficacy of the SurVeil Drug-Coated Balloon (DCB) for treatment of subjects with symptomatic peripheral artery disease (PAD) due to stenosis of the femoral and/or popliteal arteries.

DETAILED DESCRIPTION:
TRANSCEND is a prospective, multi-center, single-blind, randomized, controlled, noninferiority clinical trial. The trial will randomize approximately 446 subjects with symptomatic PAD due to stenoses of the femoral and/or popliteal arteries. Subjects meeting eligibility criteria will be randomized 1:1 to treatment with either the SurVeil DCB or the IN.PACT Admiral DCB, and followed for 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years.
* Subject has target limb Rutherford classification 2, 3 or 4.
* Subject has provided written informed consent and is willing to comply with study follow-up requirements.
* De novo lesion(s) or non-stented restenotic lesion(s) occurring >90 days after prior plain old balloon (POBA) angioplasty or >180 days after prior DCB treatment.
* Target lesion location starts ≥10 mm below the common femoral bifurcation and terminates distally at or above the end of the P1 segment of the popliteal artery.
* Target vessel diameter ≥4 mm and ≤7 mm.
* Target lesion must have angiographic evidence of ≥70% stenosis by operator visual estimate.
* Chronic total occlusions may be included only after successful, uncomplicated wire crossing of target lesion via an anterograde approach and without the use of subintimal dissection techniques.
* Target lesion must be ≤180 mm in length (one long lesion or multiple serial lesions) by operator visual estimate. Note: combination lesions must have a total lesion length of ≤180 mm by visual estimate and be separated by ≤30 mm.
* Target lesion is located at least 30 mm from any stent, if target vessel was previously stented.
* Successful, uncomplicated (without use of a crossing device) wire crossing of target lesion. Successful crossing of the target lesion occurs when the tip of the guide wire is distal to the target lesion without the occurrence of flow-limiting dissection or perforation and is judged by visual inspection to be within the true lumen.
* After pre-dilatation, the target lesion is ≤70% residual stenosis, absence of a flow limiting dissection and treatable with available device matrix.
* A patent inflow artery free from significant stenosis (≥50% stenosis) as confirmed by angiography.
* At least one patent native outflow artery to the ankle or foot, free from significant stenosis (≥50% stenosis) as confirmed by angiography.

Exclusion Criteria:

* Subject has acute limb ischemia.
* Subject underwent percutaneous transluminal angioplasty (PTA) of the target limb using plain old balloon angioplasty (POBA) or a stent within the previous 90 days.
* Subject underwent any lower extremity percutaneous treatment using a paclitaxel-eluting stent or a DCB within the previous 90 days.
* Subject underwent PTA of the target lesion using a DCB within the previous 180 days.
* Subject has had prior vascular intervention in the contralateral limb within 14 days before the planned study index procedure or subject has planned vascular intervention in the contralateral limb within 30 days after the index procedure.
* Subject is pregnant, breast-feeding or intends to become pregnant during the time of the study.
* Subject has life expectancy less than 2 years.
* Subject has a known allergy to contrast medium that cannot be adequately pre-medicated.
* Subject is allergic to ALL antiplatelet treatments.
* Subject has impaired renal function (i.e. serum creatinine level ≥2.5 mg/dL).
* Subject is dialysis dependent.
* Subject is receiving immunosuppressant therapy.
* Subject has known or suspected active infection at the time of the index procedure.
* Subject has platelet count <100,000/mm3 or >700,000/mm3.
* Subject has history of gastrointestinal hemorrhage requiring a transfusion within 3 months prior to the study procedure.
* Subject is diagnosed with coagulopathy that precludes treatment with systemic anticoagulation and/or dual antiplatelet therapy (DAPT).
* Subject has history of stroke within the past 90 days.
* Subject has a history of myocardial infarction within the past 30 days.
* Subject is unable to tolerate blood transfusions because of religious beliefs or other reasons.
* Subject is incarcerated, mentally incompetent, or abusing drugs or alcohol.
* Subject is participating in another investigational drug or medical device study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints from this study, or subject is planning to participate in such studies prior to the completion of this study.
* Subject has had any major (e.g. cardiac, peripheral, abdominal) surgical procedure or intervention unrelated to this study within 30 days prior to the index procedure or has planned major surgical procedure or intervention within 30 days of the index procedure.
* Subject had previous bypass surgery of the target lesion.
* Subject had previous treatment of the target vessel with thrombolysis or surgery.
* Subject is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol.
* Target lesion has severe calcification (as defined by the PARC classification of calcification).
* Target lesion involves an aneurysm or is adjacent to an aneurysm (within 5 mm).
* Target lesion requires treatment with alternative therapy such as stenting, laser, atherectomy, cryoplasty, brachytherapy, re-entry devices, or subintimal dissection techniques.
* Significant target vessel tortuosity or other parameters prohibiting access to the target lesion.
* Presence of thrombus in the target vessel.
* Iliac inflow disease requiring treatment, unless the iliac artery disease is successfully treated first during the index procedure. Success is defined as ≤30% residual diameter stenosis without death or major complications.
* Presence of an aortic, iliac or femoral artificial graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2024-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Lankenau Heart Group; Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital; Marianne Brodmann, MD, Principal Investigator — Medical University Graz, Department of Internal Medicine
Locations (63):
- United States (50):
  - Cardiovascular Associates of the Southeast, Birmingham, Alabama
  - Cardiology Associates, Foley, Alabama
  - Dignity Health, Gilbert, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - Mission Cardiovascular Research Institute, Fremont, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Advent Health Ocala/MediQuest Research Group LLC (formerly FL Hospital /Munroe), Ocala, Florida
  - Piedmont Heart Insitute, Atlanta, Georgia
  - Emory University Hospital (Clifton), Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Advocate Health, Naperville, Illinois
  - Prairie Education (PERC), Springfield, Illinois
  - St Vincent Heart (Research Department), Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Endovascular Technologies, LLC, Bossier City, Louisiana
  - Cardiovascular Associates Research, Covington, Louisiana
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - Northern Michigan Hospital, Petoskey, Michigan
  - North Memorial Hospital, Robbinsdale, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Mercy Hospital, Springfield, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Virtua Medical Group, P.A., Cherry Hill, New Jersey
  - St. Michael's Hospital, Newark, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Columbia University Medical Center/NYPH, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - Moses Cone-LeBauer, Greensboro, North Carolina
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - North Ohio Heart Center, Elyria, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Providence Heart and Vascular, Portland, Oregon
  - Capital Area Research, Camp Hill, Pennsylvania
  - Bryn Mawr Hospital - Main Line Health System (Einstein), Philadelphia, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Ballad Health System, Kingsport, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - St. David's Heart & Vascular PLLC dba Austin Heart, Austin, Texas
  - Houston Cardiovascular Association, Houston, Texas
  - North Dallas Research Associates, McKinney, Texas
- Prince of Wales Private Hostpital, Randwick, Australia
- Institution Medizinische Universitat, Graz, Austria
- Belgium (2):
  - AZ Sint Blasius, Dendermonde
  - UZ GENT, Ghent
- Czechia (2):
  - FN u sv. Anny v Brně a LF MU (Centrum cévních onemocnění II. chirurgická klinika), Brno
  - Vitkovicka Nemocnice Ostrava Vítkovická nemocnice, a.s.,, Ostrava
- Germany (4):
  - Herz Zentrum Bad Krozingen Südring, Bad Krozingen
  - SRH Klinikum KarlsbadLangensteinbach, Karlsbad
  - Universitätsklinikum Leipzig, Leipzig
  - REGIOMED-KLINIKEN GmbH, Sonneberg
- Aou Careggi University Hospital, Florence, Italy
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Laird JR, Schneider PA, Tepe G, Brodmann M, Zeller T, Metzger C, Krishnan P, Scheinert D, Micari A, Cohen DJ, Wang H, Hasenbank MS, Jaff MR; IN.PACT SFA Trial Investigators. Durability of Treatment Effect Using a Drug-Coated Balloon for Femoropopliteal Lesions: 24-Month Results of IN.PACT SFA. J Am Coll Cardiol. 2015 Dec 1;66(21):2329-2338. doi: 10.1016/j.jacc.2015.09.063. Epub 2015 Oct 14. PMID 26476467
- [Background] Rosenfield K, Jaff MR, White CJ, Rocha-Singh K, Mena-Hurtado C, Metzger DC, Brodmann M, Pilger E, Zeller T, Krishnan P, Gammon R, Muller-Hulsbeck S, Nehler MR, Benenati JF, Scheinert D; LEVANT 2 Investigators. Trial of a Paclitaxel-Coated Balloon for Femoropopliteal Artery Disease. N Engl J Med. 2015 Jul 9;373(2):145-53. doi: 10.1056/NEJMoa1406235. Epub 2015 Jun 24. PMID 26106946
- [Background] Patel MR, Conte MS, Cutlip DE, Dib N, Geraghty P, Gray W, Hiatt WR, Ho M, Ikeda K, Ikeno F, Jaff MR, Jones WS, Kawahara M, Lookstein RA, Mehran R, Misra S, Norgren L, Olin JW, Povsic TJ, Rosenfield K, Rundback J, Shamoun F, Tcheng J, Tsai TT, Suzuki Y, Vranckx P, Wiechmann BN, White CJ, Yokoi H, Krucoff MW. Evaluation and treatment of patients with lower extremity peripheral artery disease: consensus definitions from Peripheral Academic Research Consortium (PARC). J Am Coll Cardiol. 2015 Mar 10;65(9):931-41. doi: 10.1016/j.jacc.2014.12.036. PMID 25744011
- [Derived] Brodmann M, Gray WA, Schneider PA, Kurzmann-Guetl K, Schweiger L, Zeller T, Thieme M, Kilaru S, Bachinsky WB, Feldman RL, Holden A, Varcoe RL, Lansky AJ, Rosenfield K; TRANSCEND Study Investigators. Editor's Choice - Results of SurVeil Versus IN.PACT Admiral Paclitaxel Coated Balloons in Femoropopliteal Arteries: 24 Month Outcomes of the Randomised TRANSCEND Study. Eur J Vasc Endovasc Surg. 2025 Mar;69(3):452-462. doi: 10.1016/j.ejvs.2024.11.351. Epub 2024 Nov 29. PMID 39615582
- [Derived] Elmariah S, Ansel GM, Brodmann M, Doros G, Fuller S, Gray WA, Pinto DS, Rosenfield KA, Mauri L. Design and rationale of a randomized noninferiority trial to evaluate the SurVeil drug-coated balloon in subjects with stenotic lesions of the femoropopliteal artery - the TRANSCEND study. Am Heart J. 2019 Mar;209:88-96. doi: 10.1016/j.ahj.2018.12.012. Epub 2018 Dec 28. PMID 30685679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with symptomatic PAD presenting for percutaneous revascularization of stenosed femoral and/or popliteal arteries (either de novo lesions or non-stented restenotic lesions >90 days from prior POBA angioplasty or >180 days from prior DCB treatment) will be screened according to the protocol inclusion and exclusion criteria. Enrolled subjects who have met all the clinical inclusion criteria and none of the clinical exclusion criteria will then be screened for angiographic criteria.
Pre-assignment Details: Subjects screened via angiographic assessment to confirm remaining study eligibility prior to randomization. Subjects not meeting criteria were considered screen failures and exited from the study.
Period: Randomization
Arm/Group | Surmodics SurVeil DCB | Medtronic IN.PACT Admiral DCB
Started | 222 | 224
Completed | 222 | 224
Not Completed | 0 | 0
Period: 1-Month Visit (30 Days, - 2 to +15 Days)
Arm/Group | Surmodics SurVeil DCB | Medtronic IN.PACT Admiral DCB
Started | 222 | 224
Completed | 215 | 224
Not Completed | 7 | 0
Period: 6-Month Visit (180 Days +/- 30 Days)
Arm/Group | Surmodics SurVeil DCB | Medtronic IN.PACT Admiral DCB
Started | 215 | 224
Completed | 209 | 223
Not Completed | 6 | 1
Period: 12-Month Visit (365 Days +/- 30 Days)
Arm/Group | Surmodics SurVeil DCB | Medtronic IN.PACT Admiral DCB
Started | 209 | 223
Completed | 198 | 214
Not Completed | 11 | 9
Period: 24-Month Visit (730 Days +/- 60 Days)
Arm/Group | Surmodics SurVeil DCB | Medtronic IN.PACT Admiral DCB
Started | 198 | 214
Completed | 184 | 200
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surmodics SurVeil DCB | Medtronic IN.PACT Admiral DCB | Total
Number analyzed (Participants) | 222 | 224 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.4) | 67.4 (9.3) | 68.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 82 | 165
  Male | 139 | 142 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 212 | 216 | 428
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 21 | 44
  White | 191 | 199 | 390
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Primary Lesion Patency Though 12 Months
Description: Composite of freedom from clinically-driven target lesion revascularization (TLR) and binary restenosis (restenosis defined as duplex ultrasound [DUS] peak systolic velocity ratio [PSVR] ≥2.4 or ≥50% stenosis as assessed by independent angiographic and DUS core labs) through 12 months post-index procedure.
Time Frame: 12 months
Population: The primary analysis of the primary effectiveness endpoint was carried out on all randomized participants. For participants missing primary effectiveness endpoint status (48 for SurVeil DCB and 31 for IN.PACT Admiral DCB), a logistic regression model was used for multiple imputation with pre-specified baseline variables as model predictors.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Groups:
- SurVeil DCB: Participants randomized to receive treatment with the SurVeil DCB.
- IN.PACT Admiral DCB: Participants randomized to receive treatment with the IN.PACT Admiral DCB.
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 222 | 224
percentage of participants | 82.2 [76.4 to 87.9] | 85.9 [80.8 to 91.0]
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; The SurVeil DCB will be declared noninferior to IN.PACT Admiral DCB with respect to efficacy endpoint if the null hypothesis of inferiority is rejected at a one-sided significance level of 0.025; Test type: Non-Inferiority — 15.0% is the absolute noninferiority margin (50% of the difference in primary patency rate between IN.PACT Admiral DCB and PTA); p = 0.0029, Farrington-Manning test — P-value is derived from one-sided Farrington-Manning test with noninferiority margin of 15% and a one-sided significance level of 0.025; Difference in percentage = -3.7, 97.5% CI 1-sided [lower limit -11.7] — For subjects missing primary effectiveness endpoint status, a logistic regression model was used for multiple imputation with pre-specified baseline variables as model predictors

2. Primary Outcome: Safety Composite of Freedom From Death, Amputation, and Target Vessel Revascularization (TVR)
Description: Composite of freedom from device- and procedure-related death through 30 days post-index procedure and freedom from major target limb amputation (above the ankle) and clinically-driven TVR through 12 months post-index procedure.
Time Frame: 12 months
Population: Multiple Imputation was carried out on Intention-to-Treat (ITT) subjects. For subjects missing primary safety endpoint status, a logistic regression model was used for multiple imputation with pre-specified baseline variables as model predictors.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 222 | 224
percentage of participants | 91.8 [88.0 to 95.6] | 89.8 [85.8 to 93.8]
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; The SurVeil DCB will be declared noninferior to IN.PACT Admiral DCB with respect to safety endpoint if the null hypothesis of inferiority is rejected at a one-sided significance level of 0.025; Test type: Non-Inferiority — 10.0% is the absolute noninferiority margin (50% of the difference in primary safety endpoint rate between IN.PACT Admiral DCB and PTA); p < .0001, Farrington-Manning test — P-value is derived from one-sided Farrington-Manning test with noninferiority margin of 10% and a one-sided significance level of 0.025; Difference in percentage = 2.0, 97.5% CI 1-sided [lower limit -4.1] — For subjects missing primary safety endpoint status, a logistic regression model was used for multiple imputation with pre-specified baseline variables as model predictors

3. Secondary Outcome: Proportion of Participants With Device Success
Description: Defined as successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below rated burst pressure, and achievement of <50% residual stenosis of the target lesion (by core lab-assessed quantitative angiography [QA]) without flow-limiting arterial dissection (≥ 50% residual stenosis or dissection grade E or F) using only the study device.
Time Frame: Day 0
Population: Intention-to-Treat (ITT) Analysis Population with quantitative angiography completed by an angiography core lab.
Measure: Count of Participants; unit: Participants
Groups:
- Surmodics SurVeil DCB: Participants randomized to receive treatment with the SurVeil DCB.
Arm/Group | Surmodics SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 216 | 222
Participants | 199 | 208
Statistical Analysis 1: Comparison: Surmodics SurVeil DCB vs IN.PACT Admiral DCB; The incidence estimates will be reported along with a p-value from a two-sided Fisher's exact test comparing the SurVeil and the IN.PACT Admiral groups; Test type: Superiority; p = 0.579, Fisher Exact — P-value is derived from two-sided Fisher's exact test

4. Secondary Outcome: Proportion of Participants With Technical Success
Description: Defined as achievement of a final residual diameter stenosis of <50% (by core lab-assessed QA) without flow-limiting arterial dissection at the end of the procedure.
Time Frame: Day 0
Population: Intention-to-Treat (ITT) Analysis Population with quantitative angiography completed by an angiography core lab.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 217 | 223
Participants | 217 | 223
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; The incidence estimates will be reported along with a two-sided Fisher's exact test comparing the SurVeil and the IN.PACT Admiral groups; Test type: Superiority; p = 1.00, Fisher Exact — Both arms demonstrated 100% success, therefore, Fisher's exact test does not provide a p-value, but we populated it with a p-value of 1.00 to indicate no difference between arms

5. Secondary Outcome: Proportion of Participants With Procedure Success
Description: Defined as evidence of both acute technical success and absence of Peripheral Academic Research Consortium major adverse events (PARC MAEs; e.g., death, stroke, myocardial infarction, acute onset of limb ischemia, index bypass graft or treated segment thrombosis, and or need for urgent/emergent vascular surgery) within 72 hours of the index procedure.
Time Frame: 72 hours
Population: Intention-to-Treat (ITT) Analysis Population
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 218 | 223
Participants | 217 | 222
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 1.000, Fisher Exact — P-value is derived from two-sided Fisher's exact test

6. Secondary Outcome: Freedom From All-cause Death, Major Target Limb Amputation and TVR Through 30 Days
Description: Proportion of participation free of all-cause death, major target limb amputation and TVR through 30 days. All clinical endpoints adjudications by independent, blinded CEC.
Time Frame: 30 days
Population: Intent-to-Treat Analysis Population with assessments/follow-up completed through 30 days and/or subjects who experienced the endpoint (or any of its components) were included in the analysis (i.e., counted in the denominator).
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 218 | 223
Participants | 217 | 223
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.494, Fisher Exact — P-value is derived from two-sided Fisher's exact test

7. Secondary Outcome: Proportion of Participants With Primary Lesion Patency
Description: Primary patency through 24 months (only if both the primary safety and efficacy hypotheses of noninferiority are met).
Time Frame: 24 months
Population: The analysis was carried out on ITT subjects with available data (i.e., subjects who experienced CD-TLR through 790 days and/or binary restenosis through 24 months, or had at least 670 days of follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 154 | 181
Participants | 100 | 121
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; The objective is to assess whether the primary patency rate of subjects in the SurVeil DCB group is noninferior to that of the IN.PACT Admiral DCB group:; Test type: Non-Inferiority — The Farrington and Manning test for noninferiority of proportions at a one-sided significance level of 0.025; p = 0.0059, Farrington-Manning test — [p-value comment as in outcome 1, analysis 1]; Difference in percentage = -1.9, 97.5% CI 1-sided [lower limit -12.1]

8. Secondary Outcome: Proportion of Participants With Target Vessel Patency
Description: Defined as freedom from clinically-driven target vessel revascularization (TVR) and binary restenosis (restenosis defined as DUS PSVR ≥2.4 or ≥50% stenosis as assessed by independent angiographic and DUS core labs) within 12 and 24 months.
Time Frame: 12 months, 24 months
Population: Intention-to-Treat (ITT) analysis population with available data (i.e., subjects who experienced CD-TLR through 790 days and/or binary restenosis through 24 months, or had at least 670 days of follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 180 | 203
Participants
  Target Vessel Patency at 12-Months | 143 | 165
  Target Vessel Patency at 24-Months: number analyzed (Participants) | 163 | 187
  Target Vessel Patency at 24-Months | 102 | 118
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; The main analysis of the secondary endpoints will be carried out using the ITT analysis set; Test type: Superiority — Target Vessel Patency for SurVeil DCB vs. Target Vessel Patency for IN.PACT DCB at 12 months; p = 0.699, Fisher Exact — 12-Month P-Value
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; The main analysis of the secondary endpoints will be carried out using the ITT analysis set; Test type: Superiority — Target Vessel Patency for SurVeil DCB vs. Target Vessel Patency for IN.PACT DCB at 24 months; p = 1.0, Fisher Exact — 24-Month P-Value

9. Secondary Outcome: Proportion of Participants With Sustained Clinical Improvement
Description: Defined as freedom from major target limb amputation, TVR and worsening target limb Rutherford class, within 6, 12, and 24 months.
Time Frame: 6 months, 12 months, 24 months
Population: Intent-to-Treat analysis population consisting of participants either experiencing the event within the period or who have adequate follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 195 | 208
Participants
  6-Months | 158 | 172
  12-Months: number analyzed (Participants) | 184 | 204
  12-Months | 121 | 142
  24-Months: number analyzed (Participants) | 164 | 186
  24-Months | 93 | 111
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.699, Fisher Exact — 6-Month P-Value
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.447, Fisher Exact — 12-Month P-Value
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.589, Fisher Exact — 24-Month P-Value

10. Secondary Outcome: Proportion of Participants With a Clinically-Driven Target Lesion Revascularization (TLR)
Description: Includes participants experiencing a clinically-driven target lesion revascularization event as reported by sites and adjudicated by an independent CEC.
Time Frame: 6 months, 12 months, 24 months
Population: Intent-to-Treat analysis population consisting of participants either experiencing the event within the period (e.g., 30 days for 1-month time point, 180 days for 6-month time point, 365 days for 12-month time point, 730 days for 24-month time point) or who have adequate follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 209 | 222
Participants
  Clinically-driven TLR at 6-Months | 3 | 3
  Clinically-driven TLR at 12-Months: number analyzed (Participants) | 201 | 217
  Clinically-driven TLR at 12-Months | 11 | 10
  Clinically-driven TLR at 24-Months: number analyzed (Participants) | 186 | 205
  Clinically-driven TLR at 24-Months | 27 | 24
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact — P-Value at 6-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.823, Fisher Exact — P-Value at 12-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.454, Fisher Exact — P-Value at 24-Months

11. Secondary Outcome: Proportion of Participants With a Historical Major Adverse Events (MAEs)
Description: MAEs defined as composite of all-cause death, clinically-driven TLR, major target limb amputation, or thrombosis at the target lesion, within 6, 12, 24 months.
Time Frame: 6 months, 12 months, 24 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 212 | 223
Participants
  Historical MAEs at 6-Months | 6 | 4
  Historical MAEs at 12-Months: number analyzed (Participants) | 206 | 221
  Historical MAEs at 12-Months | 17 | 17
  Historical MAEs at 24-Months: number analyzed (Participants) | 201 | 218
  Historical MAEs at 24-Months | 43 | 39
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.535, Fisher Exact — P-Value at 6-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.860, Fisher Exact — P-Value at 12-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.390, Fisher Exact — P-Value at 24-Months

12. Secondary Outcome: Proportion of Participants With a Major Target Limb Amputation
Description: Major target limb amputation within 6, 12, 24 months as reported by site and adjudicated by CEC.
Time Frame: 6 months, 12 months, 24 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 208 | 222
Participants
  Major Target Limb Amputation at 6-Months | 0 | 0
  Major Target Limb Amputation at 12-Months: number analyzed (Participants) | 199 | 217
  Major Target Limb Amputation at 12-Months | 0 | 0
  Major Target Limb Amputation at 24-Months: number analyzed (Participants) | 183 | 205
  Major Target Limb Amputation at 24-Months | 0 | 1
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.00, Fisher Exact — Both arms demonstrated 0 amputations at 6 months. Fisher's Exact test does not provide a p-value, but we populated it with a p-value of 1.00 to indicate no difference between arms
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.00, Fisher Exact — Both arms demonstrated 0 amputations at 12 months. Fisher's Exact test does not provide a p-value, but we populated it with a p-value of 1.00 to indicate no difference between arms
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact — P-Value at 24-Months

13. Secondary Outcome: Proportion of Participants With a Thrombosis at the Target Lesion.
Description: Thrombosis at target lesion within 6, 12, 24 months as reported by the site and adjudicated by the CEC.
Time Frame: 6 months, 12 months, 24 months
Population: Intent-to-Treat analysis population consisting of participants either experiencing the event within the period (e.g., 30 days for 1-month time point, 180 days for 6-month time point, 365 days for 12-month time point, 760 days for 24-month time point) or who have adequate follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 208 | 222
Participants
  Thrombosis at Target Lesion at 6-Months | 0 | 0
  Thrombosis at Target Lesion at 12-Months: number analyzed (Participants) | 199 | 217
  Thrombosis at Target Lesion at 12-Months | 0 | 0
  Thrombosis at Target Lesion at 24-Months: number analyzed (Participants) | 183 | 205
  Thrombosis at Target Lesion at 24-Months | 1 | 0
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.472, Fisher Exact — P-Value at 24-Months

14. Secondary Outcome: Change in Target Limb Rutherford Class
Description: Change in target limb Rutherford class from Baseline (BL) to 1, 6, 12, and 24 months.
  Rutherford classification criteria categorize the severity of chronic limb ischemia based on a clinical description of symptoms and pre-defined objective criteria.
  Possible scores range from 0 to 6 (with lower scores representing a better outcome) with scores defined as follows:
  0 - Asymptomatic - no hemodynamically significant occlusive disease
  1. - Mild claudication
  2. - Moderate claudication
  3. - Severe claudication
  4. - Ischemic rest pain
  5. - Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia
  6. - Major tissue loss, extending above transmetatarsal) with all scores defined as follows:
  Change = 1-Month scores - BL scores; 6-Month scores - BL scores; 12-Month scores - BL scores; 24-Month scores - BL scores
Time Frame: Baseline, 1 month, 6 months, 12 months, and 24 months
Population: Analysis of the secondary endpoint includes the Intention-to-Treat analysis population for whom Rutherford classification was available at the respective timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 210 | 220
Participants
  Change in Rutherford Classification from Baseline to 1-Month: Grade ≥+3 Markedly improved | 101 | 90
  Change in Rutherford Classification from Baseline to 1-Month: Grade +2 Moderately improved | 63 | 78
  Change in Rutherford Classification from Baseline to 1-Month: Grade +1 Mildly improved | 28 | 29
  Change in Rutherford Classification from Baseline to 1-Month: No change | 16 | 20
  Change in Rutherford Classification from Baseline to 1-Month: Grade -1 Mildly worsening | 1 | 2
  Change in Rutherford Classification from Baseline to 1-Month: Grade -2 Moderately worsening | 0 | 0
  Change in Rutherford Classification from Baseline to 1-Month: Grade ≤-3 Markedly worsening | 1 | 1
  Change in Rutherford Classification from Baseline to 6-Months: number analyzed (Participants) | 195 | 209
  Change in Rutherford Classification from Baseline to 6-Months: Grade ≥+3 Markedly improved | 101 | 95
  Change in Rutherford Classification from Baseline to 6-Months: Grade +2 Moderately improved | 65 | 70
  Change in Rutherford Classification from Baseline to 6-Months: Grade +1 Mildly improved | 15 | 30
  Change in Rutherford Classification from Baseline to 6-Months: No change | 11 | 12
  Change in Rutherford Classification from Baseline to 6-Months: Grade -1 Mildly worsening | 1 | 2
  Change in Rutherford Classification from Baseline to 6-Months: Grade -2 Moderately worsening | 1 | 0
  Change in Rutherford Classification from Baseline to 6-Months: Grade ≤-3 Markedly worsening | 1 | 0
  Change in Rutherford Classification from Baseline to 12-Months: number analyzed (Participants) | 183 | 204
  Change in Rutherford Classification from Baseline to 12-Months: Grade ≥+3 Markedly improved | 82 | 74
  Change in Rutherford Classification from Baseline to 12-Months: Grade +2 Moderately improved | 50 | 76
  Change in Rutherford Classification from Baseline to 12-Months: Grade +1 Mildly improved | 28 | 33
  Change in Rutherford Classification from Baseline to 12-Months: No change | 18 | 16
  Change in Rutherford Classification from Baseline to 12-Months: Grade -1 Mildly worsening | 5 | 3
  Change in Rutherford Classification from Baseline to 12-Months: Grade -2 Moderately worsening | 0 | 2
  Change in Rutherford Classification from Baseline to 12-Months: Grade ≤-3 Markedly worsening | 0 | 0
  Change in Rutherford Classification from Baseline to 24-Months: number analyzed (Participants) | 157 | 178
  Change in Rutherford Classification from Baseline to 24-Months: Grade ≥+3 Markedly improved | 77 | 65
  Change in Rutherford Classification from Baseline to 24-Months: Grade +2 Moderately improved | 36 | 60
  Change in Rutherford Classification from Baseline to 24-Months: Grade +1 Mildly improved | 26 | 34
  Change in Rutherford Classification from Baseline to 24-Months: No change | 17 | 14
  Change in Rutherford Classification from Baseline to 24-Months: Grade -1 Mildly worsening | 1 | 4
  Change in Rutherford Classification from Baseline to 24-Months: Grade -2 Moderately worsening | 0 | 1
  Change in Rutherford Classification from Baseline to 24-Months: Grade ≤-3 Markedly worsening | 0 | 0
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.193, Wilcoxon (Mann-Whitney) — P-Value for change in Rutherford Classification from BL to 1-Month
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.140, Wilcoxon (Mann-Whitney) — P-Value for change in Rutherford Classification from BL to 6-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.372, Wilcoxon (Mann-Whitney) — P-Value for change in Rutherford Classification from BL to 12-Months
Statistical Analysis 4: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.104, Wilcoxon (Mann-Whitney) — P-Value for change in Rutherford Classification from BL to 24-Months

15. Secondary Outcome: Change in Target Limb Peripheral Academic Research Consortium (PARC) Class
Description: Change in target limb PARC class from baseline to 1, 6, 12, and 24 months.
  PARC definitions of clinical symptom classification were used to classify subject claudication at baseline and subsequent follow-up visits. PARC clinical symptom classification is used to capture information regarding lower extremity symptoms and broadly define functional limitations of patients with lower extremity peripheral artery disease (PAD).
  Possible classifications (asymptomatic=best outcome to ischemic gangrene=worst outcome) include the following:
  Asymptomatic Mild claudication/limb symptoms (no limitation in walking) Moderate claudication/limb symptoms (able to walk without stopping > 2 blocks or 200 meters or 4 minutes) Severe claudication/limb symptoms (only able to walk without stopping < 2 blocks or 200 meters or 4 minutes) Ischemic rest pain (pain in the distal limb at rest, felt to be due to limited arterial perfusion) Ischemic ulcers on distal leg Ischemic gangrene
  Change =
Time Frame: Screening, 1 month, 6 months, 12 months, and 24 months
Population: Analysis of the secondary endpoint includes the Intention-to-Treat analysis population for whom PARC clinical classification was available at the respective timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 210 | 221
Participants
  Change in PARC class from BL to 1-Month: Grade ≥+3 Markedly improved | 99 | 89
  Change in PARC class from BL to 1-Month: Grade +2 Moderately improved | 59 | 78
  Change in PARC class from BL to 1-Month: Grade +1 Mildly improved | 31 | 31
  Change in PARC class from BL to 1-Month: Grade 0 No change | 18 | 18
  Change in PARC class from BL to 1-Month: Grade -1 Mildly worsening | 2 | 4
  Change in PARC class from BL to 1-Month: Grade -2 Moderately worsening | 0 | 0
  Change in PARC class from BL to 1-Month: Grade ≤-3 Markedly worsening | 1 | 1
  Change in PARC Class from BL to 6-Months: Grade ≥+3 Markedly improved: number analyzed (Participants) | 195 | 208
  Change in PARC Class from BL to 6-Months: Grade ≥+3 Markedly improved | 99 | 92
  Change in PARC Class from BL to 6-Months: Grade +2 Moderately improved: number analyzed (Participants) | 195 | 208
  Change in PARC Class from BL to 6-Months: Grade +2 Moderately improved | 65 | 70
  Change in PARC Class from BL to 6-Months: Grade +1 Mildly improved: number analyzed (Participants) | 195 | 208
  Change in PARC Class from BL to 6-Months: Grade +1 Mildly improved | 16 | 30
  Change in PARC Class from BL to 6-Months: Grade 0 No change: number analyzed (Participants) | 195 | 208
  Change in PARC Class from BL to 6-Months: Grade 0 No change | 12 | 14
  Change in PARC Class from BL to 6-Months: Grade -1 Mildly worsening: number analyzed (Participants) | 195 | 208
  Change in PARC Class from BL to 6-Months: Grade -1 Mildly worsening | 1 | 2
  Change in PARC Class from BL to 6-Months: Grade -2 Moderately worsening: number analyzed (Participants) | 195 | 208
  Change in PARC Class from BL to 6-Months: Grade -2 Moderately worsening | 1 | 0
  Change in PARC Class from BL to 6-Months: Grade ≤-3 Markedly worsening: number analyzed (Participants) | 195 | 208
  Change in PARC Class from BL to 6-Months: Grade ≤-3 Markedly worsening | 1 | 0
  Change in PARC Class from BL to 12-Months: Grade ≥+3 Markedly improved: number analyzed (Participants) | 183 | 203
  Change in PARC Class from BL to 12-Months: Grade ≥+3 Markedly improved | 80 | 69
  Change in PARC Class from BL to 12-Months: Grade +2 Moderately improved: number analyzed (Participants) | 183 | 203
  Change in PARC Class from BL to 12-Months: Grade +2 Moderately improved | 53 | 80
  Change in PARC Class from BL to 12-Months: Grade +1 Mildly improved: number analyzed (Participants) | 183 | 203
  Change in PARC Class from BL to 12-Months: Grade +1 Mildly improved | 27 | 31
  Change in PARC Class from BL to 12-Months: Grade 0 No change: number analyzed (Participants) | 183 | 203
  Change in PARC Class from BL to 12-Months: Grade 0 No change | 17 | 17
  Change in PARC Class from BL to 12-Months: Grade -1 Mildly worsening: number analyzed (Participants) | 183 | 203
  Change in PARC Class from BL to 12-Months: Grade -1 Mildly worsening | 6 | 4
  Change in PARC Class from BL to 12-Months: Grade -2 Moderately worsening: number analyzed (Participants) | 183 | 203
  Change in PARC Class from BL to 12-Months: Grade -2 Moderately worsening | 0 | 1
  Change in PARC Class from BL to 12-Months: Grade ≤-3 Markedly worsening: number analyzed (Participants) | 183 | 203
  Change in PARC Class from BL to 12-Months: Grade ≤-3 Markedly worsening | 0 | 1
  Change in PARC Classification from BL to 24-Months: Grade ≥+3 Markedly improved: number analyzed (Participants) | 156 | 178
  Change in PARC Classification from BL to 24-Months: Grade ≥+3 Markedly improved | 73 | 63
  Change in PARC Classification from BL to 24-Months: Grade +2 Moderately improved: number analyzed (Participants) | 156 | 178
  Change in PARC Classification from BL to 24-Months: Grade +2 Moderately improved | 37 | 62
  Change in PARC Classification from BL to 24-Months: Grade +1 Mildly improved: number analyzed (Participants) | 156 | 178
  Change in PARC Classification from BL to 24-Months: Grade +1 Mildly improved | 25 | 33
  Change in PARC Classification from BL to 24-Months: Grade 0 No change: number analyzed (Participants) | 156 | 178
  Change in PARC Classification from BL to 24-Months: Grade 0 No change | 19 | 14
  Change in PARC Classification from BL to 24-Months: Grade -1 Mildly worsening: number analyzed (Participants) | 156 | 178
  Change in PARC Classification from BL to 24-Months: Grade -1 Mildly worsening | 2 | 5
  Change in PARC Classification from BL to 24-Months: Grade -2 Moderately worsening: number analyzed (Participants) | 156 | 178
  Change in PARC Classification from BL to 24-Months: Grade -2 Moderately worsening | 0 | 1
  Change in PARC Classification from BL to 24-Months: Grade ≤-3 Markedly worsening: number analyzed (Participants) | 156 | 178
  Change in PARC Classification from BL to 24-Months: Grade ≤-3 Markedly worsening | 0 | 0
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.320, Wilcoxon (Mann-Whitney) — P-Value for change in PARC from BL to 1-Month
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.132, Wilcoxon (Mann-Whitney) — P-Value for change in PARC from BL to 6-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.248, Wilcoxon (Mann-Whitney) — P-Value for change in PARC from BL to 12-Months
Statistical Analysis 4: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.194, Wilcoxon (Mann-Whitney) — P-Value for change in PARC from BL to 24-Months

16. Secondary Outcome: Decrease in Target Limb Resting Ankle Brachial Index (ABI) or Toe Brachial Index (TBI)
Description: Decrease in target limb resting ABI or TBI ≥0.15 from baseline to 6, 12, and 24 months.
  Ankle-brachial index (ABI) is the ratio of the systolic blood pressure (SBP) measured at the ankle to that measured at the brachial artery.
  Toe brachial index (TBI) is the ratio of SBP measured at the toe to that measured at the brachial artery.
  if ABI could not be assessed, TBI could be used.
Time Frame: Screening, 6 months, 12 months, and 24 months
Population: Analysis of the secondary endpoint includes the Intention-to-Treat analysis population for whom the ABI or TBI was available at the respective timepoint. Worsening of ABI was defined as a decrease in ABI ≥0.15 from baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 183 | 199
Participants
  BL to 6-Months: Decrease in Resting Target Limb ABI ≥0.15 | 6 | 8
  BL to 6-Months: Decrease in Resting Target Limb TBI ≥0.15: number analyzed (Participants) | 9 | 10
  BL to 6-Months: Decrease in Resting Target Limb TBI ≥0.15 | 0 | 0
  BL to 12-Months: Decrease in Resting Target Limb ABI ≥0.15: number analyzed (Participants) | 174 | 189
  BL to 12-Months: Decrease in Resting Target Limb ABI ≥0.15 | 15 | 6
  BL to 12-Months: Decrease in Resting Target Limb TBI ≥0.15: number analyzed (Participants) | 11 | 8
  BL to 12-Months: Decrease in Resting Target Limb TBI ≥0.15 | 2 | 1
  BL to 24-Months: Decrease in Resting Target Limb ABI ≥0.15: number analyzed (Participants) | 149 | 172
  BL to 24-Months: Decrease in Resting Target Limb ABI ≥0.15 | 9 | 15
  BL to 24-Months: Decrease in Resting Target Limb TBI ≥0.15: number analyzed (Participants) | 12 | 12
  BL to 24-Months: Decrease in Resting Target Limb TBI ≥0.15 | 1 | 1
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.789, Fisher Exact — P-Value for Decrease in Resting Target Limb ABI ≥0.15: BL to 6-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.041, Fisher Exact — P-Value for Decrease in Resting Target Limb ABI ≥0.15: BL to 12-Months
Statistical Analysis 4: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact — P-Value for Decrease in Resting Target Limb TBI ≥0.15: BL to 12-Months
Statistical Analysis 5: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.401, Fisher Exact — P-Value for Decrease in Resting Target Limb ABI ≥0.15: BL to 24-Months
Statistical Analysis 6: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact — P-Value for Decrease in Resting Target Limb TBI ≥0.15: BL to 24-Months

17. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ)
Description: Walking Impairment Questionnaire is a validated tool that has 4 domains (Walking Impairment, Walking Distance, Walking Speed, and Stair Climbing), each scored as a percent ranging from 0 (representing the inability to perform any of the tasks) to 100 (representing no difficulty with any of the tasks). A positive change in a score indicates an improvement.
Time Frame: Screening, 1 month, 12 months, and 24 months
Population: Intention-to-Treat population for whom Walking Impairment Questionnaire information was available from Baseline to each respective time point.
  An increase in a WIQ score signifies improvement.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 204 | 219
score on a scale
  Change from BL to 1-Month: Walking Impairment Score | 50.0 [25.0 to 75.0] | 50.0 [25.0 to 75.0]
  Change from BL to 1-Month: Walking Distance Score: number analyzed (Participants) | 203 | 218
  Change from BL to 1-Month: Walking Distance Score | 37.6 [1.8 to 70.3] | 23.4 [0.1 to 65.0]
  Change from BL to 1-Month: Walking Speed Score: number analyzed (Participants) | 198 | 215
  Change from BL to 1-Month: Walking Speed Score | 15.2 [0.0 to 43.5] | 15.2 [0.0 to 34.8]
  Change from BL to 1-Month: Stair Climbing Score: number analyzed (Participants) | 200 | 217
  Change from BL to 1-Month: Stair Climbing Score | 20.8 [0.0 to 54.2] | 12.5 [0.0 to 45.8]
  Change from BL to 12-Months: Walking Impairment Score: number analyzed (Participants) | 181 | 205
  Change from BL to 12-Months: Walking Impairment Score | 25.0 [0.0 to 75.0] | 50.0 [25.0 to 75.0]
  Change from BL to 12-Months: Walking Distance Score: number analyzed (Participants) | 181 | 204
  Change from BL to 12-Months: Walking Distance Score | 26.3 [0.0 to 62.9] | 27.7 [1.1 to 66.9]
  Change from BL to 12-Months: Walking Speed Score: number analyzed (Participants) | 178 | 205
  Change from BL to 12-Months: Walking Speed Score | 17.4 [0.0 to 43.5] | 17.4 [0.0 to 43.5]
  Change from BL to 12-Months: Stair Climbing Score: number analyzed (Participants) | 180 | 205
  Change from BL to 12-Months: Stair Climbing Score | 20.8 [-4.2 to 47.9] | 20.8 [0.0 to 54.2]
  Change from BL to 24-Months: Walking Impairment Score: number analyzed (Participants) | 162 | 185
  Change from BL to 24-Months: Walking Impairment Score | 50.0 [0.0 to 75.0] | 50.0 [0.0 to 75.0]
  Change from BL to 24-Months: Walking Distance Score: number analyzed (Participants) | 162 | 184
  Change from BL to 24-Months: Walking Distance Score | 26.8 [-0.4 to 61.8] | 27.6 [0.0 to 65.1]
  Change from BL to 24-Months: Walking Speed Score: number analyzed (Participants) | 160 | 184
  Change from BL to 24-Months: Walking Speed Score | 10.9 [-6.0 to 40.8] | 12.0 [-3.8 to 39.1]
  Change from BL to 24-Months: Stair Climbing Score: number analyzed (Participants) | 161 | 185
  Change from BL to 24-Months: Stair Climbing Score | 20.8 [-4.2 to 45.8] | 16.7 [0.0 to 45.8]
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Other; p = 0.995, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 1-Month: Walking Impairment Score
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.158, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 1-month: Walking distance score
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.695, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 1-month: Walking speed score
Statistical Analysis 4: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.086, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 1-Month: Stair Climbing Score
Statistical Analysis 5: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.331, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 12-Months: Walking Impairment Score
Statistical Analysis 6: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.580, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 12-Months: Walking Distance Score
Statistical Analysis 7: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.563, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 12-Months: Walking Speed Score
Statistical Analysis 8: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.270, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 12-Months: Stair Climbing Score
Statistical Analysis 9: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.869, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 24-Months: Walking Impairment Score
Statistical Analysis 10: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.837, Wilcoxon (Mann-Whitney) — P-value for change in WIQ from BL to 24-Months: Walking Distance Score
Statistical Analysis 11: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.674, Wilcoxon (Mann-Whitney) — P-value for change in WIQ for BL to 24-Months: Walking Speed Score
Statistical Analysis 12: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.563, Wilcoxon (Mann-Whitney) — P-value for change in WIQ for BL to 24-Months: Stair Climbing Score

18. Secondary Outcome: Change in 6-Minute Walk Test (6MWT)
Description: Change in 6MWT from baseline to 12 and 24 months.
Time Frame: Screening, 12 months, and 24 months
Population: Intention-to-Treat population for whom the 6-Minute Walk Test information from Baseline to each respective time point was available.
Measure: Mean (Standard Deviation); unit: Distance walked (meters)
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 163 | 180
Distance walked (meters)
  Change from BL to 12-Months | 45.8 (118.8) | 60.7 (113.6)
  Change from BL to 24-Months: number analyzed (Participants) | 128 | 161
  Change from BL to 24-Months | 25.7 (98.8) | 52.5 (122.4)
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.237, t-test, 2 sided — P-value for change in 6MWT from BL to 12-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.040, t-test, 2 sided — P-value for change in 6MWT from BL to 24-Months

19. Secondary Outcome: Change in Peripheral Artery Questionnaire (PAQ)
Description: The PAQ consists of 7 domains including physical function, stability, symptom, treatment satisfaction, quality of life, social limitation, and summary. Scores range from 0 to 100, with a positive change indicating an improvement. Questionnaire responses include: Extremely Limited, Quite a bit Limited, Moderately Limited, Slightly Limited, Not at all Limited, Limited for other reasons or did not do the activity.
Time Frame: Screening, 1 month, 12 months, and 24 months
Population: Intention-to-Treat Analysis Population for whom the PAQ score information from baseline to each respective time point was available.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 203 | 219
score on a scale
  1-Month: Physical Function Score: number analyzed (Participants) | 178 | 196
  1-Month: Physical Function Score | 25.0 [4.2 to 58.3] | 29.2 [8.3 to 50.0]
  1-Month: Stability Score | 50.0 [0.0 to 50.0] | 50.0 [25.0 to 50.0]
  1-Month: Symptom Score | 33.3 [11.1 to 52.8] | 30.6 [8.3 to 50.0]
  1-Month: Treatment Satisfaction Score: number analyzed (Participants) | 202 | 219
  1-Month: Treatment Satisfaction Score | 0.0 [0.0 to 8.3] | 0.0 [0.0 to 16.7]
  1-Month: Quality of Life Score | 41.7 [16.7 to 58.3] | 33.3 [16.7 to 50.0]
  1-Month: Social Limitation Score: number analyzed (Participants) | 177 | 202
  1-Month: Social Limitation Score | 25.0 [8.3 to 50.0] | 25.0 [8.3 to 50.0]
  1-Month: Summary Score | 32.6 [10.4 to 52.8] | 30.2 [13.2 to 46.6]
  12-Months: Physical Function Score: number analyzed (Participants) | 161 | 178
  12-Months: Physical Function Score | 25.0 [4.2 to 45.8] | 25.0 [8.3 to 54.2]
  12-Months: Stability Score: number analyzed (Participants) | 180 | 205
  12-Months: Stability Score | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 25.0]
  12-Months: Symptom Score: number analyzed (Participants) | 180 | 205
  12-Months: Symptom Score | 27.8 [8.3 to 47.2] | 30.6 [5.6 to 52.8]
  12-Months: Treatment Satisfaction Score: number analyzed (Participants) | 179 | 205
  12-Months: Treatment Satisfaction Score | 0.0 [-8.3 to 8.3] | 0.0 [0.0 to 8.3]
  12-Months: Quality of Life Score: number analyzed (Participants) | 180 | 205
  12-Months: Quality of Life Score | 33.3 [16.7 to 58.3] | 33.3 [8.3 to 58.3]
  12-Months: Social Limitation Score: number analyzed (Participants) | 162 | 183
  12-Months: Social Limitation Score | 25.0 [8.3 to 50.0] | 25.0 [8.3 to 58.3]
  12-Months: Summary Score: number analyzed (Participants) | 180 | 205
  12-Months: Summary Score | 29.7 [13.4 to 49.1] | 30.3 [9.7 to 52.8]
  24-Months: Physical Function Score: number analyzed (Participants) | 139 | 163
  24-Months: Physical Function Score | 25.0 [4.2 to 50.0] | 29.2 [4.2 to 54.2]
  24-Month: Stability Score: number analyzed (Participants) | 163 | 185
  24-Month: Stability Score | 0.0 [0.0 to 25.0] | 0.0 [0.0 to 25.0]
  24-Months: Symptom Score: number analyzed (Participants) | 163 | 185
  24-Months: Symptom Score | 27.8 [11.1 to 50.0] | 33.3 [13.9 to 52.8]
  24-Months: Treatment Satisfaction Score: number analyzed (Participants) | 162 | 185
  24-Months: Treatment Satisfaction Score | 0.0 [0.0 to 8.3] | 0.0 [0.0 to 8.3]
  24-Months: Quality of Life Score: number analyzed (Participants) | 163 | 185
  24-Months: Quality of Life Score | 41.7 [16.7 to 58.3] | 33.3 [16.7 to 58.3]
  24-Months: Social Limitation Score: number analyzed (Participants) | 145 | 160
  24-Months: Social Limitation Score | 25.0 [8.3 to 50.0] | 25.0 [8.3 to 50.0]
  24-Months: Summary Score: number analyzed (Participants) | 163 | 185
  24-Months: Summary Score | 29.9 [12.5 to 48.3] | 28.5 [13.9 to 49.9]
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.772, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 1-Month: Physical Function Score
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.930, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 1-Month: Stability Score
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.546, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 1-Month: Symptom Score
Statistical Analysis 4: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.621, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 1-Month: Treatment Satisfaction Score
Statistical Analysis 5: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.133, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 1-Month: Quality of Life Score
Statistical Analysis 6: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.592, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 1-Month: Social Limitation Score
Statistical Analysis 7: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.601, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 1-Month: Summary Score
Statistical Analysis 8: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.185, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months: Physical Function Score
Statistical Analysis 9: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.856, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months: Stability Score
Statistical Analysis 10: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.541, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months: Symptom Score
Statistical Analysis 11: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.731, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months: Treatment Satisfaction Score
Statistical Analysis 12: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.696, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months: Quality of Life Score
Statistical Analysis 13: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.716, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months: Social Limitation Score
Statistical Analysis 14: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.797, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months: Summary Score
Statistical Analysis 15: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.290, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 24-Months: Physical Function Score
Statistical Analysis 16: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.473, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 24-Months: Stability Score
Statistical Analysis 17: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.278, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 24-Months: Symptom Score
Statistical Analysis 18: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.974, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 24-Months: Treatment Satisfaction Score
Statistical Analysis 19: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.266, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 24-Months: Quality of Life Score
Statistical Analysis 20: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.656, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 24-Months: Social Limitation Score
Statistical Analysis 21: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.959, Wilcoxon (Mann-Whitney) — P-value for change in PAQ from BL to 12-Months:Summary Score

20. Secondary Outcome: Proportion of Participants With a Clinically-Driven Target Lesion Revascularization (TLR)
Description: as for outcome 10
Time Frame: 36 months, 48 months, 60 months
Population: Intent-to-Treat analysis population consisting of participants either experiencing the event within the period (e.g., 1095 days for 36-month time point, 1460 days for 48-month time point,1825 days for 60-month time point) or who have adequate follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 179 | 195
Participants
  Clinically-driven TLR at 36-Months | 36 | 39
  Clinically-driven TLR at 486-Months: number analyzed (Participants) | 170 | 188
  Clinically-driven TLR at 486-Months | 42 | 48
  Clinically-driven TLR at 60-Months: number analyzed (Participants) | 161 | 179
  Clinically-driven TLR at 60-Months | 44 | 50
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact — P-Value at 36-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.903, Fisher Exact — P-Value at 48-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact — P-Value at 60-Months

21. Secondary Outcome: Proportion of Participants With a Historical Major Adverse Events (MAEs)
Description: MAEs defined as composite of all-cause death, clinically-driven TLR, major target limb amputation, or thrombosis at the target lesion within 36, 48, and 60 months.
Time Frame: 36 months, 48 months, 60 months
Population: Intent-to-Treat analysis population consisting of participants either experiencing the event within the period (e.g., 1095 days for 36-month time point, 1460 days for 48--month time point, 1825 days for 60-month time point) or who have adequate follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 198 | 214
Participants
  Historical MAEs at 36-Months | 56 | 62
  Historical MAEs at 48-Months: number analyzed (Participants) | 197 | 214
  Historical MAEs at 48-Months | 69 | 75
  Historical MAEs at 60-Months: number analyzed (Participants) | 194 | 211
  Historical MAEs at 60-Months | 79 | 83
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.913, Fisher Exact; P-Value at 36-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact; P-Value at 48-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.839, Fisher Exact — P-Value at 60-Months

22. Secondary Outcome: Proportion of Participants With a Major Target Limb Amputation
Description: Major target limb amputation within 36, 48, and 60 months as reported by site and adjudicated by CEC.
Time Frame: 36 months, 48 months, 60 months
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 174 | 191
Participants
  Major Target Limb Amputation at 36-Months | 0 | 1
  Major Target Limb Amputation at 48-Months: number analyzed (Participants) | 163 | 182
  Major Target Limb Amputation at 48-Months | 0 | 2
  Major Target Limb Amputation at 60-Months: number analyzed (Participants) | 150 | 172
  Major Target Limb Amputation at 60-Months | 0 | 3
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 1.0, Fisher Exact — P-Value at 36-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.5, Fisher Exact; P-Value at 48-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.251, Fisher Exact; P-Value at 60-Months

23. Secondary Outcome: Proportion of Participants With a Thrombosis at the Target Lesion
Description: Thrombosis at target lesions within 36, 48, and 60 months as reported by the site and adjudicated by the CEC.
Time Frame: 36 months, 48 months, 60 months
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | SurVeil DCB | IN.PACT Admiral DCB
Number analyzed (Participants) | 175 | 191
Participants
  Thrombosis at Target Lesion at 36-Months | 1 | 0
  Thrombosis at Target Lesion at 48-Months: number analyzed (Participants) | 164 | 182
  Thrombosis at Target Lesion at 48-Months | 2 | 1
  Thrombosis at Target Lesion at 60-Months: number analyzed (Participants) | 152 | 172
  Thrombosis at Target Lesion at 60-Months | 3 | 1
Statistical Analysis 1: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.478, Fisher Exact — P-Value at 36-Months
Statistical Analysis 2: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.605, Fisher Exact — P-Value at 48-Months
Statistical Analysis 3: Comparison: SurVeil DCB vs IN.PACT Admiral DCB; Test type: Superiority; p = 0.345, Fisher Exact — P-Value at 60-Months

ADVERSE EVENTS:
Time Frame: Enrollment through 60-months
Arm/Group | Surmodics SurVeil DCB | Medtronic IN.PACT Admiral DCB
All-Cause Mortality (participants affected / at risk) | 41/222 | 37/224
Serious Adverse Events (participants affected / at risk) | 166/222 | 162/224
Other Adverse Events (participants affected / at risk) | 159/222 | 170/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surmodics SurVeil DCB (N=222) | Medtronic IN.PACT Admiral DCB (N=224)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 15 (19) | 23 (29)
Angina pectoris (Cardiac disorders) | 9 (10) | 4 (4)
Angina unstable (Cardiac disorders) | 4 (4) | 3 (4)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 9 (12) | 9 (12)
Atrial flutter (Cardiac disorders) | 3 (4) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac arrest (Cardiac disorders) | 8 (8) | 4 (4)
Cardiac failure (Cardiac disorders) | 4 (4) | 3 (4)
Cardiac failure acute (Cardiac disorders) | 6 (14) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 9 (9) | 8 (10)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 9 (10) | 13 (18)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 4 (5)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (4)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Urachal abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (6) | 7 (9)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site discharge (General disorders) | 2 (2) | 0 (0)
Catheter site haematoma (General disorders) | 3 (3) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1)
Drug withdrawal syndrome (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 3 (3) | 1 (1)
Mass (General disorders) | 0 (0) | 1 (1)
Necrosis (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (8) | 4 (5)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Vascular stent occlusion (General disorders) | 2 (3) | 5 (5)
Vascular stent restenosis (General disorders) | 3 (5) | 7 (7)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 5 (6) | 2 (2)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 6 (6) | 10 (10)
Cystitis (Infections and infestations) | 0 (0) | 3 (4)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Haematoma infection (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (14) | 9 (11)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 7 (8) | 7 (8)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (6) | 5 (5)
Vascular access site infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 3 (3) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 15 (17) | 11 (18)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (4) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
5q minus syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 6 (6) | 6 (7)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 5 (5)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 2 (3)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (3)
Epidural lipomatosis (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 4 (4)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 8 (9) | 3 (3)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 3 (3)
Device malfunction (Product Issues) | 1 (2) | 2 (2)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 15 (18) | 12 (13)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (2) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital erosion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (10)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 6 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 7 (8)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 2 (3)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (2)
Aortic intramural haematoma (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 4 (4)
Arterial spasm (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 3 (4)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 2 (3) | 7 (8)
Ischaemic limb pain (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 3 (3)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 10 (13) | 10 (12)
Peripheral artery aneurysm (Vascular disorders) | 2 (4) | 2 (2)
Peripheral artery dissection (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 23 (35) | 22 (34)
Peripheral artery stenosis (Vascular disorders) | 44 (64) | 35 (50)
Peripheral embolism (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 11 (15) | 7 (11)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 3 (3)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Subclavian steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (2) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surmodics SurVeil DCB (N=222) | Medtronic IN.PACT Admiral DCB (N=224)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 6 (6) | 6 (6)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 3 (3)
Coronary artery disease (Cardiac disorders) | 2 (2) | 4 (4)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 2 (3)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (4) | 6 (8)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eyelid dermatochalasis (Eye disorders) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Ocular vascular disorder (Eye disorders) | 1 (1) | 0 (0)
Retinal drusen (Eye disorders) | 1 (1) | 0 (0)
Retinopathy hypertensive (Eye disorders) | 1 (1) | 0 (0)
Vitreous adhesions (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 5 (5)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (6) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal angioedema (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Reactive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Uvulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (5)
Asthenia (General disorders) | 2 (2) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 8 (8) | 8 (8)
Catheter site haemorrhage (General disorders) | 2 (2) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 3 (3)
Chest pain (General disorders) | 1 (1) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 3 (3)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Implant site extravasation (General disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 8 (12) | 6 (8)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 6 (7) | 16 (19)
Peripheral swelling (General disorders) | 2 (2) | 8 (8)
Vascular stent occlusion (General disorders) | 0 (0) | 1 (1)
Vascular stent restenosis (General disorders) | 2 (2) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 6 (6)
Cellulitis (Infections and infestations) | 3 (3) | 4 (4)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 12 (12) | 6 (6)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 3 (3)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 3 (3) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 11 (12) | 7 (9)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 5 (6)
Epidural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Laceration (Injury, poisoning and procedural complications) | 2 (3) | 4 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 7 (8) | 16 (17)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood glucose abnormal (Investigations) | 2 (2) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2) | 1 (1)
Heart sounds abnormal (Investigations) | 0 (0) | 1 (1)
Lipoprotein (a) increased (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Ultrasound Doppler abnormal (Investigations) | 0 (0) | 1 (1)
Ultrasound scan abnormal (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 10 (11)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (8)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (21) | 15 (17)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (7) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 7 (8)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalomalacia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 5 (5) | 4 (4)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 3 (3)
Radiculopathy (Nervous system disorders) | 1 (3) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (6) | 2 (2)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular acidosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5)
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 8 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis atrophic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (6)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Aortic dilatation (Vascular disorders) | 1 (1) | 0 (0)
Aortic occlusion (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 3 (3) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (2) | 0 (0)
Arterial insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis Moenckeberg-type (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Atheroembolism (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Femoral artery dissection (Vascular disorders) | 18 (18) | 22 (22)
Haematoma (Vascular disorders) | 2 (2) | 3 (3)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 11 (12) | 9 (10)
Hypertensive crisis (Vascular disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 8 (8) | 1 (1)
Intermittent claudication (Vascular disorders) | 19 (21) | 14 (16)
Lower limb artery perforation (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 7 (7) | 6 (6)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 7 (8) | 10 (11)
Peripheral artery stenosis (Vascular disorders) | 30 (37) | 34 (41)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 1 (1)
Secondary hypertension (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 0 (0) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03241459/Prot_SAP_000.pdf